CLINICAL TRIAL: NCT00458588
Title: Adolescent Diet, Hormones and Breast Cancer Susceptibility
Brief Title: Long-Term Effect of Adolescent Diet on Hormones and Breast Cancer Risk in Women Previously Enrolled in the Dietary Intervention Study in Children
Status: Completed | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000538232; R01CA104670 (NIH); P30CA006927 (NIH); FCCC-9305; FCCC-IRB-05-843
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Absorptiometry, Photon; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Other: physiologic testing
Other: questionnaire administration
Procedure: breast imaging study
Procedure: dual x-ray absorptometry
Procedure: evaluation of cancer risk factors
Procedure: magnetic resonance imaging

SUMMARY:
RATIONALE: The amount and type of fat in the diet may affect hormone levels, bone mineral density, and breast density later in life. This may affect the risk of developing breast cancer. Learning about the long-term effects of diet on hormone levels, bone mineral density, and breast density may help the study of breast cancer in the future.

PURPOSE: This clinical trial is studying the long-term effect of adolescent diet on hormones and breast cancer risk in women previously enrolled in the Dietary Intervention Study in Children.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the long-term effect of the Dietary Intervention Study in Children (DISC) to lower total fat and saturated fat intake during adolescence on serum progesterone levels in young women previously enrolled in the DISC study.

Secondary

* Determine the long-term effect of the DISC intervention on serum estradiol levels in these women.
* Determine the long-term effect of the DISC intervention on bone mineral density in these women.
* Determine the long-term effect of the DISC intervention on breast density in these women.
* Determine the long-term effect of the DISC intervention on the prevalence of metabolic syndrome in these women.

OUTLINE: This is a multicenter study.

Patients undergo fasting blood collection on day 1 for assessment of serum hormones (progesterone, estradiol), lipids, lipoproteins, and fasting glucose. Patients also undergo blood pressure, height, weight, and waist circumference measurements. Patient then receive a snack and complete the Modifiable Activity questionnaire, Center for Epidemiological Studies Depression Scale short form, Spielberger State-Trait Anxiety Inventory, and Dietary Intervention Study in Children Medical History questionnaire (including demographics, medical history, menstrual history, medications, reproductive history, dietary supplements, alcohol and tobacco use, and family history of cancer). Patients also undergo dual-energy x-ray absorptiometry (DEXA) and MRI to measure bone and breast density. Patients complete an in-person 24-hour dietary recall using the Nutrition Data System for Research on day 1 and via telephone once in weeks 2 and 3.

Day 1 is scheduled during the patient's luteal phase of menstrual cycle. After completion of study, patients contact the clinic to report start of next menses.

PROJECTED ACCRUAL: A total of 301 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Previously enrolled on a clinical trial titled, "Dietary Intervention Study in Children"

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent females
Sampling Method: Probability Sample
Enrollment: 301 (Estimated)
Dates: Start 2006-09 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Mean serum progesterone level in women not using hormonal contraceptives | Day 1 of treatment

SECONDARY OUTCOMES:
Luteal phase serum estradiol level in women not using hormonal contraceptives | Day 1 of treatment
Bone mineral density of women who are not pregnant | Day 1 of treatment
Breast density of women who are not pregnant | Day 1 of treatment
Prevalence of metabolic syndrome | Day 1 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Dorgan, PhD, MPH, Study Chair — Fox Chase Cancer Center
Locations (10):
- United States (10):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Maryland Medical Research Institute, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - UMDNJ University Hospital, Newark, New Jersey
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Jung S, Goloubeva O, Hylton N, Klifa C, LeBlanc E, Shepherd J, Snetselaar L, Van Horn L, Dorgan JF. Intake of dietary carbohydrates in early adulthood and adolescence and breast density among young women. Cancer Causes Control. 2018 Jul;29(7):631-642. doi: 10.1007/s10552-018-1040-1. Epub 2018 May 25. PMID 29802491
- [Derived] Bertrand KA, Baer HJ, Orav EJ, Klifa C, Kumar A, Hylton NM, LeBlanc ES, Snetselaar LG, Van Horn L, Dorgan JF. Early Life Body Fatness, Serum Anti-Mullerian Hormone, and Breast Density in Young Adult Women. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1151-7. doi: 10.1158/1055-9965.EPI-16-0185. Epub 2016 May 9. PMID 27197299
- [Derived] Bertrand KA, Baer HJ, Orav EJ, Klifa C, Shepherd JA, Van Horn L, Snetselaar L, Stevens VJ, Hylton NM, Dorgan JF. Body fatness during childhood and adolescence and breast density in young women: a prospective analysis. Breast Cancer Res. 2015 Jul 16;17(1):95. doi: 10.1186/s13058-015-0601-4. PMID 26174168
- [Derived] Jung S, Egleston BL, Chandler DW, Van Horn L, Hylton NM, Klifa CC, Lasser NL, LeBlanc ES, Paris K, Shepherd JA, Snetselaar LG, Stanczyk FZ, Stevens VJ, Dorgan JF. Adolescent endogenous sex hormones and breast density in early adulthood. Breast Cancer Res. 2015 Jun 4;17(1):77. doi: 10.1186/s13058-015-0581-4. PMID 26041651
- [Derived] Jung S, Stanczyk FZ, Egleston BL, Snetselaar LG, Stevens VJ, Shepherd JA, Van Horn L, LeBlanc ES, Paris K, Klifa C, Dorgan JF. Endogenous sex hormones and breast density in young women. Cancer Epidemiol Biomarkers Prev. 2015 Feb;24(2):369-78. doi: 10.1158/1055-9965.EPI-14-0939. Epub 2014 Nov 4. PMID 25371447
- [Derived] Dorgan JF, Liu L, Barton BA, Deshmukh S, Snetselaar LG, Van Horn L, Stevens VJ, Robson AM, Lasser NL, Himes JH, Shepherd JA, Pourfarzib R, Pettee Gabriel K, Kriska A, Kwiterovich PO Jr. Adolescent diet and metabolic syndrome in young women: results of the Dietary Intervention Study in Children (DISC) follow-up study. J Clin Endocrinol Metab. 2011 Dec;96(12):E1999-2008. doi: 10.1210/jc.2010-2726. Epub 2011 Oct 12. PMID 21994964